CLINICAL TRIAL: NCT05837533
Title: Multicenter Study to Evaluate the Impact of a Systematized Communication Model to Increase the Knowledge of Breast Cancer Patients About Their Disease
Brief Title: Multicenter Study to Evaluate a Systematized Communication Model for Breast Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medicos e Investigadores en la Lucha contra el Cancer de Mama (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Double | Purpose: Other
Other Study IDs: EC-COMUNICACION
Record Dates: First submitted 2023-04-19; First posted 2023-05-01 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer Stage IV; Breast Cancer Metastatic; Communication
MeSH Terms: conditions — Breast Neoplasms; Communication

STUDY DESIGN:
Intervention Model Description: During the first half of the study, patients will be assigned to the control group where they will receive information through their usual care from their oncologist during their medical consultation. In the second half of the study, patients will be assigned to the intervention group where they will receive information through the communication model used by their oncologist during their medical consultation. In this way, the contamination of the control group with attention corresponding to the systematized communication model under study will be avoided.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will not be informed whether they will be allocated to the control or intervention group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): Patients will receive information about their diagnosis, treatment and/or prognosis through the systematic communication model under study used by their oncologist during their medical consultation.
  Interventions: Other: Communication model
- Control group (No Intervention): Patients will receive information about their diagnosis, treatment and/or prognosis through their usual care provided by their oncologist during their medical consultation.

INTERVENTIONS:
Other: Communication model — During the medical consultation of each patient assigned to the intervention group, the oncologist will use the systematic communication model for patients with metastatic breast cancer. For this, the oncologist will follow the conversation guide for patients with metastatic breast cancer, which will allow directing the conversation towards information about the patient's diagnosis, treatment and prognosis. The guide consists of a series of steps and questions to be asked to the patient in order to explore her understanding of her disease and her information preferences, as well as to facilitate the oncologist providing said information to the patient. The responses to each item in the guide will be electronically documented by the oncologist.
  Arms: Intervention group

SUMMARY:
Both in Mexico and in the world, breast cancer is the most common malignancy in women. It is estimated that in 2020, 28.2% of the new cancer cases reported in our country correspond to breast cancer, which translates to 30,000 new cases. In addition, it is relevant to mention that approximately 12% of Mexican patients are diagnosed with stage IV breast cancer and it is estimated that 20-30% of women with early stage cancer will have a distant recurrence of the disease. Thus, about 40% of patients will find themselves in a metastatic stage at some point in their breast cancer journey.

Various studies, including Mexico, report that only half of patients with metastatic breast cancer are aware that their disease is not curable, 31% say they are not sure, and 17% think it is curable. Likewise, 58% considered that they did not have enough knowledge to actively participate in conversations about their therapeutic options, which means that 40% reported difficulty talking about treatments with their doctors. This has shown that there are suboptimal levels of knowledge information on curability, treatment objectives and prognosis of their condition in patients with metastatic breast cancer. This lack of understanding is alarming given that a general understanding of the disease is crucial for informed decision making and adherence to cancer treatment.

Due to these alarming results, we seek to recruit women ≥18 years of age who are candidates to start first- or second-line treatment for de novo or recurrent metastatic breast cancer from various hospital centers in the country with public and private coverage, including Hospital Zambrano Hellion TecSalud as coordinating center in Nuevo León. The objective will be to evaluate whether a systematized communication model for patients with metastatic breast cancer allows increasing knowledge about the non-curative nature of treatment, compared to usual care.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of de novo or recurrent metastatic breast cancer
* Candidate to start the first or second line of treatment for metastatic breast cancer

Exclusion Criteria:

* Receipt of a line of treatment for metastatic breast cancer posterior to the second line

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-05-17 (Actual); Primary Completion 2024-11-16 (Actual); Study Completion 2024-11-16 (Actual)

PRIMARY OUTCOMES:
Patient understanding | 7 days
  Evaluate whether a systematic communication model for patients with metastatic breast cancer increases patients' understanding about the non-curative nature of treatment, compared to usual care. Understanding will be measured with the "Knowledge questionnaire" consisting of the Prognosis and Treatment Perceptions Questionnaire (PTPQ) questions, which explore patients' beliefs about their possibility of cure and the main objective of their treatment, their perception of the importance and usefulness of knowing their prognosis, their information preferences, as well as their satisfaction with the quality of the information received. Additionally, the research group developed specific questions that are of interest for this study to assess participants' perception of the usefulness of the information received through the systematic communication model, as well as their use of the information materials provided and their degree of satisfaction with them.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Zambrano Hellion, San Pedro Garza García, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: No